CLINICAL TRIAL: NCT02510833
Title: Home Therapeutic Exercises Oriented for People With Parkinson's Disease: Impact on the Disease and Quality of Life
Brief Title: Effects of Home Therapeutic Exercises Oriented for Patients With Parkinson's Disease
Acronym: HTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, IHANA THAÍS GUERRA DE OLIVEIRA GONDIM, IHANA THAÍS GUERRA DE OLIVEIRA GONDIM, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE- 38511314000005208
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Physical Therapy Modalities; Quality of Life; Self Care
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuing Intervention Group (Experimental)
  Interventions: Behavioral: Exercises oriented, manual and monitoring by phone
- Control Group (Active Comparator)
  Interventions: Behavioral: Exercises oriented, manual and without monitoring by phone

INTERVENTIONS:
Behavioral: Exercises oriented, manual and monitoring by phone — Individual meeting to guide therapeutic exercises (stretching, mobility, balance and strength), manual with these exercises for support in practice at home and weekly monitoring by phone. Patients will be oriented to do exercises three times per week for twelve weeks.
  Arms: Continuing Intervention Group
Behavioral: Exercises oriented, manual and without monitoring by phone — Lectures (optatives) about therapeutic exercises (stretching, mobility, balance and strength) in days of medical consultation, manual with these exercises for support in practice at home, without weekly monitoring by phone. Patients will be oriented to do exercises three times per week for twelve weeks.
  Arms: Control Group

SUMMARY:
Parkinson's disease (PD), neurodegenerative and common from 50 to 60 years, is characterized by rigidity, bradykinesia and resting tremor that can interfere in the quality of life. To maintain or improve this, there is the physiotherapy. Problems in access, such as walking and financial difficulties, make home exercises target of interest. The study aims to assess the impact of a program of home therapeutic exercises, with individualized approach and remote monitoring by physical therapist, about signs and symptoms of Parkinson's disease and quality of life. This is a randomized controlled clinical trial, conducted at the Program Pró-Parkinson of the Clinics Hospital, Federal University of Pernambuco, Neurology Clinic. Will be included people of both sexes (50 years) with idiopathic PD, stages 1-3 in Hoehn & Yahr original; non-institutionalized and independent walking. It will be applied before and after 12 weeks of intervention (period ON of medication): Survey about Knowledge, Attitudes and Practice; Questionnaire of Accession; Unified Scale Evaluation of Parkinson's disease (UPDRS) - subscales II and III; and Parkinson's Disease Questionnaire 39 (PDQ-39). Participants will be randomized into two groups: Group continued intervention (GIC) and control group (CG). The GIC will have an meeting with individualized approach (physical therapist, patient and companion) for guidance on home physical therapy exercises, using the Manual Pró-Parkinson, then the participant will receive the manual with stretching exercises, mobility, balance and strength, which will lead to your home as a way to guide their activities; and receive weekly follow-up by phone calls (to remember the exercises, answer questions and encourage the continued practice). GC may be attend presentations on home exercises of the Pro-Parkinson's manual in the days of your query and have the same manual without remote follow-up by phone calls, usual service procedure. Exercises are oriented to be performed three times a week for 12 weeks and under the effect of anti-Parkinson medication. This study will contribute new evidence on the effects of a rehabilitation program available and inexpensive based on home exercises.

DETAILED DESCRIPTION:
Type of Study:

Randomized controlled clinical trial.

Hypothesis:

Program-oriented home therapeutic exercises with individualized approach and weekly monitoring of the physical therapist contributes to the improvement of signs and symptoms of Parkinson's disease and quality of life.

Primary objective:

To evaluate the impact of home therapeutic exercises oriented in people with Parkinson's disease.

Secondary objective:

* To investigate the knowledge, attitudes and practice about home therapeutic exercises oriented in the study population;
* Identify adhesion and barriers related to exercise program;
* Evaluate the impact of home-based therapeutic exercise about daily activities, motor exploration and the quality of life in Parkinson's disease.

Proposed Methodology:

Participants will be informed of the nature and purpose of the study. Then those who meet the eligibility criteria and wish to participate, sign the Consent Agreement and Informed (IC). The study will be conducted in the Pró-Parkinson Program at the Hospital das Clinicas, Federal University of Pernambuco (UFPE), Neurology Clinic, between December/ 2014 to September/2015. Will be applicable before and after 12 weeks of intervention ( medication ON period): Survey about Knowledge, Attitudes and Practice; Questionnaire of Accession; Unified Scale Evaluation of Parkinson's disease (UPDRS) - subscales II and III; and Parkinson's Disease Questionnaire 39 (PDQ-39). Participants will be randomized into two groups: Group continued intervention (GIC) and control group (CG). GIC- Initially, a physiotherapist, member of the Pró-Parkinson Program and responsible for this research, guide and train the individual patient and his companion about physiotherapy exercises present in an illustrative manual of the Pro-Parkinson. Also, there are lectures about the therapeutic exercises in in medical consultation day. The exercises should be performed in his home three times a week (every other day) with a maximum duration of 60 minutes each session for 12 weeks and always under the influence of anti-Parkinsonian medications (ON period of medication). After the meeting, receive the manual, if not yet available, and a daily exercises. In the diary, the participant or caregiver should write down the exercises, reporting the day, time, held all or not and difficulties for subsequent control of the responsible researcher. Participants will receive weekly calls from physiotherapist at the agreed time with the participant and / or caregiver, to remind them of the exercises, answer questions and encourage them to continue the practice. It is emphasized that if the participant and caregiver this are not able to write in the diary, the data will be questioned by the researcher in his weekly phone call, without prejudice to the control. Physiotherapist phone numbers will be available for participants in the daily exercises. GC- participants and accompanying persons may attend the lectures of the service (including the Physical Therapy) and have the same manual, without the subsequent weekly follow-up phone calls, usual service procedure. The lectures take place every Wednesday in day consultation, two meetings / month for the physiotherapy team. These have a maximum duration of 40 minutes in which patients and caregivers are instructed and trained to do the manual physical therapy exercises his home three times a week with a maximum duration of 60 minutes each session and always under the influence anti-Parkinsonian drugs (ON period of the medication). At the end of the talks, the manual is available. The lectures are given by physiotherapists, properly trained, the Pro-Parkinson Program members. The Pro-Parkinson manual, distributed in the program since 2012, covers chapters with exercises and guidelines of medical areas, physiotherapy, speech therapy, occupational therapy and dentistry. The physiotherapy section (page 10-21) includes stretching exercises, mobility, balance and strength, plus the guidelines. It has general instructions for the exercises; the sequence describing the same, self-explanatory illustrations and the number of sets and reps / maintenance time to be realized. All exercises are designed so they could be carried out independently and safely in the patient's home. Patients will be instructed to make them with clothes that let free knees and sneakers or shoes (if there jump up to 2 cm) that are attached to the ankle. The exercises will be supervised by the patient or caregiver, own if necessary.

Risks:

With regard to the questionnaires, there may be the risk of embarrassment. To minimize the same, the data collection will be held individually and enabling environment for data confidentiality. If refuses to answer any question, no insistence, as well as any damage to the participant. Pain, muscle discomfort or fatigue may occur during and after the exercises, however, the patient will be advised to discontinue the exercises try a case considered unbearable pain. To minimize these risks, the whole exercise program will be guided to be held in range of motion and pain-free intensity for the safety. During the exercises, you can also change the cardiorespiratory parameters such as blood pressure and respiratory rate. In an attempt to minimize risk, will not participate in the study those who submit changes in blood pressure levels and heart rate and respiratory considered beyond normal.

Benefits:

The direction of this study will bring direct benefits to patients attending the service in order to be a population with few resources to finance a rehabilitation treatment, or with little or no access to such services as with patients in the state . This diagnosis of the study population are described in Coriolanos et al. (2013) that describing the epidemiological profile of patients with PD at HC/UFPE. Moreover, the results will contribute to evidence-based therapeutic practice and the literary collection, fostering new studies.

Data Analysis Methodology:

All study collections will be held at Pró-Parkinson Program at the Hospital das Clinicas, Federal University of Pernambuco (UFPE), Neurology Clinic, and each variable will be evaluated by the responsible employees and physiotherapist, who will undergo a period of training. Outcomes will be analyzed using statistical software SPSS version 16.0 (SPSS Inc, Chicago, IL, USA). To verify the normality of the sample, the Shapiro-Wilk test is used. Upon proof of normality, the results before and after the intervention will be compared within groups, paired analysis, by means of the Wilcoxon test and intergroup, independent analysis, using the Mann-Whitney test. To analyze the results of the Survey CAP and Adhesion, the descriptive statistics from the frequency calculations will be made, high-low, median, mean, standard deviation. The significance level is 0.05 on all analyses. Datas and images through photographs will be stored on the personal computer of responsible physical therapist and counselor, and there are two copies on CD compact disc/DVD. The responsibility of confidentiality of data is the responsible physiotherapist.

Sample Size in Brazil: 28 (14 in the intervention group and 14 for control). To carry out the sample size calculation, the investigators used the statistical program PASS (Power Analysis and Sample Size), version 2005. After simulations, the investigators chose a minimum sample size of 14 patients in the control group and 14 for the intervention group, totaling 28 patients. This number is capable of detecting, with a 82% test power and 5% significance level, a reduction of 3 points in the PDQ-39 scale and UPDRS-Motor for the intervention group compared with no reduction for the control group, using a one-tailed parametric or non-parametric test for independent samples, considering the standard deviation of the reduction on the order of 3 points to the two groups. For all calculations, the mean and standard deviation parameters were expected based on studies Lun et al. (2005), Dereli and Yaliman (2010), Navarro-Peternella and Marcon (2012), as well as clinical experience Pró-Parkinson.

ELIGIBILITY:
Inclusion Criteria:

* People female and male; not institutionalized; aged between 50 and 80 years; diagnosed with idiopathic PD attested by the service neurologist in mild to moderate stages (classified from 1 to 3) in accordance with the original version of the scale of Hoehn & Yahr (HOEHN & Yahr, 1967); independent gait (without assistance)..

Exclusion Criteria:

* Those with cognitive impairment identified by the Mini Mental State Examination (MMSE) (Folstein & MC HUGH, 1975), whose cutoff point for illiterate individuals will be 18/19 and for individuals with schooling will be 24/25 (LOURENCO & VERAS, 2006 ); other neurological disorders, orthopedic limiting or unstable cardiopulmonary associated; with any medical contraindication to exercise or musculoskeletal and do physical therapy.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Unified Scale Evaluation of Parkinson's disease (UPDRS) | 3 months
  Standard evaluation to measure the signs and symptoms in practice and clinical research in PD. It consists of 42 items divided into four subscales: I- mentation, behavior and mood; II activities of daily living (ADLs); III motor operation and IV complications of drug therapy. For this study will be used only subscales II and III, with a view to clinical evaluation with a focus on activities of daily living and motor operation. The score for each item ranges from 0 to 4, and the maximum value indicates greater commitment by the disease.
Parkinson's Disease Questionnaire 39 (PDQ-39) | 3 months
  The PDQ-39 is a specific tool to assess quality of life in PD. Comprises 39 items divided into eight dimensions: mobility, activities of daily living (ADLs), emotional well-being, stigma, social support, cognition, communication and physical discomfort, where scores range from 0-100, with the higher, the worse the perception of quality of life.

SECONDARY OUTCOMES:
Survey about Knowledge, Attitudes and Practice (CAP) | 3 months
  It can be adapted to different contexts aimed at strategic planning of health promotion interventions. Prepared by the research team, will address issues relating to knowledge, attitudes and practices on a manual physical therapy exercises. Knowledge is considered adequate when the person know the exercise of the Pro-Parkinson's manual; name at least two physical therapy properly and respond to the exercises serve to "treat the disease," "improve health", "to take care" and / or "to do at home." With regard to the attitude, it will be deemed adequate if the person think you should do the physical therapy exercises at home and this is necessary. Since the practice is considered adequate when the person responds that makes manual physical therapy exercises at home, at least three days a week and practiced for the last time "this week" or "last week".
Questionnaire on Barriers identification for Accession | 3 months
  Prepared by the research team, the questionnaire will identify the barriers to entry into the program. For this, the lifting of the following data will be made: if the patient can understand how to do the exercises during physical therapy lecture; you can not understand the exercises and what their motives; presents difficulties in performing the manual physical therapy exercises at home and what their motives.

CONTACTS AND LOCATIONS:
Overall Officials: IHANA GONDIM, Principal Investigator — Universidade Federal de Pernambuco

REFERENCES:
- [Background] CORIOLANO MGWS et al. Perfil epidemiológico dos pacientes com doença de parkinson do Hospital das Clínicas da Universidade Federal de Pernambuco. Neurobiologia, 76 (1-2) jan./jun., 2013. DERELI EE, YALIMAN A. Comparison of the effects of a physiotherapist-supervised exercise programme and a self-supervised exercise programme on quality of life in patients with Parkinson's disease. Clin Rehabil. 2010;24(4):352-62. LUN, V. et al. Comparison of the effects of a self-supervised home exercise program with a physiotherapist-supervised exercise program on the motor symptoms of Parkinson's disease. Mov Dis, v. 20, n. 8, p. 971-5, 2005. NAVARRO-PETERNELLA, F. M.; MARCON, S. S. Qualidade de vida de indivíduos com Parkinson e sua relação com tempo de evolução e gravidade da doença. Rev. Latino-Am. Enfermagem, v. 20, n. 2, 2012.